CLINICAL TRIAL: NCT00160706
Title: A Phase III Multi-national, Multi-centre, Open Label, Safety Study to Assess the Safety of Re-exposure After a Variable Interval and Subsequent Chronic Therapy With the Humanised Anti-TNF PEG Conjugate CDP870 400 mg sc, (Dosed at Weeks 0, 2 and 4 Then Every 4 Weeks), in the Treatment of Patients With Active Crohn's Disease Who Have Previously Been Withdrawn From Studies CDP870-031 or CDP870-032 Due to an Exacerbation of Crohn's Disease.
Brief Title: A follow-on Safety Study in Subjects With Crohn's Disease Who Have Previously Been Withdrawn From the Double-blind Study CDP870-031 [NCT00152490] or CDP870-032 [NCT00152425] Due to an Exacerbation of Crohn's Disease
Acronym: PRECiSE 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C87034; 2005-002623-13 (EudraCT Number)
Expanded Access: NCT03559660 (No longer available)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2013-07-04 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2013-05

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Certolizumab Pegol (Experimental): 3-dose induction regimen of Certolizumab Pegol 400 mg at Weeks 0, 2, 4. Subsequently continue on 4-weekly treatment with Certolizumab Pegol 400 mg until Week 360.
  Interventions: Biological: Certolizumab Pegol (CDP870)

INTERVENTIONS:
Biological: Certolizumab Pegol (CDP870) — Liquid for subcutaneous injection, 200 mg/ml. 400 mg at Weeks 0, 2, 4 and thereafter every 4 weeks until Week 360.
  Up to 84 months of therapy in this study.
  Other Names: Cimzia; CDP870; CZP

SUMMARY:
A follow-on safety study in subjects with Crohn's Disease who have previously been withdrawn from the double-blind study CDP870-031 [NCT00152490] or CDP870-032 [NCT00152425] due to an exacerbation of Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Participation in either of the CDP870-031 [NCT00152490] or CDP870-032 [NCT00152425] clinical studies in which the subject completed the Week 2 assessment in CDP870-031 [NCT00152490] or the Week 6 randomization in CDP870-032 [NCT00152425] but whose Crohn's Disease was significantly worse as determined by the investigator and whose Clinical Disease Activity Index (CDAI) score at entry to this study is either (subjects may have received active or placebo treatment):

  1. At least 70 points higher then Baseline (Week 0 CDP870-031 [NCT00152490]; Week 6 CDP870 032 [NCT00152425] responders) OR
  2. Higher than Baseline (Week 0 CDP870-031 [NCT00152490]; Week 6 CDP870-032 [NCT00152425] responders) with an absolute score of at least 350 points
* Subjects must be able to understand the information provided to them and give written informed consent

Exclusion Criteria:

* Any exclusion criterion that would have prevented the subject's participation in the qualifying pivotal study (CDP870-031 [NCT00152490] or CDP870-032 [NCT00152425]), although the upper limit of 450 in the CDAI score is not applicable. In addition the criterion that excludes previous participation in a clinical trial of Certolizumab Pegol does not apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2004-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (141):
- United States (41):
  - 45102, Birmingham, Alabama
  - 45028, Huntsville, Alabama
  - 45044, Little Rock, Arkansas
  - 45095, Orange, California
  - 45101, San Francisco, California
  - 45130, Colorado Springs, Colorado
  - 45094, Gainesville, Florida
  - 45005, Hialeah, Florida
  - 45087, Miami, Florida
  - 45004, North Miami Beach, Florida
  - 45016, Chicago, Illinois
  - 45037, Indianapolis, Indiana
  - 45019, Lexington, Kentucky
  - 45033, Chevy Chase, Maryland
  - 45013, Laurel, Maryland
  - 45083, Rochester, Minnesota
  - 45108, Jefferson City, Missouri
  - 45035, Berlin, New Jersey
  - 45009, Great Neck, New York
  - 45070, New York, New York
  - 45145, Greenville, North Carolina
  - 45067, High Point, North Carolina
  - 45003, Raleigh, North Carolina
  - 45040, Winston-Salem, North Carolina
  - 45081, Cincinnati, Ohio
  - 45091, Cincinnati, Ohio
  - 45054, Dayton, Ohio
  - 45025, Mayfield Heights, Ohio
  - 45039, Oklahoma City, Oklahoma
  - 45041, Tulsa, Oklahoma
  - 45093, Hershey, Pennsylvania
  - 45113, Germantown, Tennessee
  - 45119, Nashville, Tennessee
  - 45022, Houston, Texas
  - 45073, San Antonio, Texas
  - 45139, Salt Lake City, Utah
  - 45052, South Ogden, Utah
  - 45134, Charlottesville, Virginia
  - 45078, Christiansburg, Virginia
  - 45109, Norfolk, Virginia
  - 45141, Seattle, Washington
- Australia (14):
  - 11011, Bankstown, New South Wales
  - 11005, New Lambton, New South Wales
  - 11017, Herston, Queensland
  - 11006, South Brisbane, Queensland
  - 11014, Lauceston, Tasmania
  - 11016, Ballarat, Victoria
  - 11007, Box Hill, Victoria
  - 11002, Fitzroy, Victoria
  - 11013, Frankston, Victoria
  - 11012, Parkville, Victoria
  - 11009, Adelaide
  - 11010, Fremantle
  - 11015, Garran
  - 11018, Newtown
- Austria (3):
  - 46006, Linz
  - 46003, Salzburg
  - 46002, Vienna
- 12001, Minsk, Belarus
- Belgium (3):
  - 13004, Brussels
  - 13001, Ghent
  - 13003, Leuven
- 15001, Sofia, Bulgaria
- Canada (4):
  - 16005, Winnipeg, Manitoba
  - 16014, Halifax, Nova Scotia
  - 16013, Toronto, Ontario
  - 16008, Montreal, Quebec
- Czechia (4):
  - 18006, Hradek Kralove
  - 18001, Ostrava
  - 18002, Prague
  - 18004, Prague
- Denmark (5):
  - 19004, Aalborg
  - 19009, Copenhagen
  - 19010, Herlev
  - 19007, Hvidovre
  - 19003, Vejle
- Estonia (2):
  - 20001, Tallinn
  - 20002, Tartu
- Germany (11):
  - 22002, Berlin
  - 22009, Berlin
  - 22004, Celle
  - 22019, Frankfurt
  - 22013, Göttingen
  - 22017, Hanover
  - 22015, Kiel
  - 22016, Leipzig
  - 22001, Minden
  - 22012, Munich
  - 22008, Münster
- Hungary (3):
  - 24002, Budapest
  - 24009, Pécs
  - 24011, Szekszárd
- Israel (3):
  - 26004, Beersheba
  - 26007, Haifa
  - 26005, Petha Tikva
- Italy (3):
  - 27001, Milan
  - 27004, Palermo
  - 27007, Roma
- New Zealand (5):
  - 31002, Auckland
  - 31001, Christchurch
  - 31005, Hamilton
  - 31004, Milford
  - 31003, Tauranga
- Norway (3):
  - 32005, Oslo
  - 32008, Oslo
  - 32004, Tromsø
- Poland (6):
  - 33008, Bydgoszcz
  - 33003, Gdansk
  - 33018, Lublin
  - 33013, Szczecin
  - 33007, Warsaw
  - 33009, Warsaw
- Russia (7):
  - 34017, Lipetsk
  - 34006, Moscow
  - 34016, Nizhny Novgorod
  - 34001, Saint Petersburg
  - 34005, Saint Petersburg
  - 34007, Saint Petersburg
  - 34013, Saint Petersburg
- Serbia (3):
  - 35001, Belgrade
  - 35002, Belgrade
  - 35004, Belgrade
- 36002, Singapore, Singapore
- Slovenia (2):
  - 38001, Celje
  - 38003, Ljubljana
- South Africa (12):
  - 39013, Johannesburg, Gauteng
  - 39003, Cape Town, Somerset West
  - 39016, Cape Town
  - 39018, Cape Town
  - 39012, Goodwood
  - 39010, Johannesburg
  - 39008, Midrand
  - 39004, Port Elizabeth
  - 39006, Pretoria
  - 39009, Pretoria
  - 39014, Pretoria
  - 39019, Pretoria
- 40009, Barcelona, Spain
- Ukraine (3):
  - 43008, Dniepropetrovsk
  - 43003, Lviv
  - 43006, Odesa

REFERENCES:
- [Result] Sandborn WJ, Schreiber S, Hanauer SB, Colombel JF, Bloomfield R, Lichtenstein GR; PRECiSE 4 Study Investigators. Reinduction with certolizumab pegol in patients with relapsed Crohn's disease: results from the PRECiSE 4 Study. Clin Gastroenterol Hepatol. 2010 Aug;8(8):696-702.e1. doi: 10.1016/j.cgh.2010.03.024. Epub 2010 Apr 2. PMID 20363366
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study started to enroll subjects in February 2004 in order to end up with 141 centers in 24 countries with enrolled subjects.
  Participant Flow refers to the Safety Population, including all enrolled subjects who received at least one injection of study treatment in feeder study C87031 [NCT00152490] or C87032 [NCT00152425].
Pre-assignment Details: Subjects who withdrew from feeder studies for worsening of Crohn's Disease entered study C87034. Subjects in study C87031 were eligible for entry into C87034 at any time after completing the Week 2 assessment, subjects in study C87032 at any time after completing the Week 6 randomisation.
Groups:
- Certolizumab Pegol: 3-dose induction regimen of Certolizumab Pegol 400 mg at Weeks 0, 2, 4. Subsequently continue on 4-weekly treatment with Certolizumab Pegol 400 mg until Week 360.
  Certolizumab Pegol (CDP870) : Liquid for subcutaneous injection, 200 mg/ml. 400 mg at Weeks 0, 2, 4 and thereafter every 4 weeks until Week 360.
  Up to 84 months of therapy in this study.
Period: Overall Study
Arm/Group | Certolizumab Pegol
Started | 310
Completed | 24
Not Completed | 286
Not completed — Adverse Event | 53
Not completed — Adverse Event and Other Reason | 105
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 41
Not completed — Withdrawal by Subject and Other | 12
Not completed — Physician Decision | 10
Not completed — Physician Decision and Other | 3
Not completed — Lost to Follow-up | 4
Not completed — Lost to Follow-up and Other | 1
Not completed — Lack of Efficacy | 42
Not completed — Lack of Efficacy and Other | 1
Not completed — Other Reason | 11

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Population, including all enrolled subjects who received at least one injection of study treatment in feeder study C87031 [NCT00152490] or C87032 [NCT00152425].
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 310
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 299
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179
  Male | 131
Region of Enrollment [Number; unit: participants]
  Serbia | 4
  United States | 74
  Belarus | 2
  Estonia | 5
  Slovenia | 3
  Spain | 1
  Ukraine | 3
  Austria | 7
  Russian Federation | 17
  Israel | 5
  Italy | 5
  Czech Republic | 10
  Hungary | 13
  Canada | 9
  Poland | 10
  Belgium | 8
  Singapore | 2
  Australia | 43
  Denmark | 11
  South Africa | 31
  Bulgaria | 1
  Norway | 7
  Germany | 29
  New Zealand | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With at Least One Adverse Event (AE) During the Duration of This Study CDP870-034 (up to 84 Months)
Description: An AE is defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Time Frame: Up to 84 months from Study Entry (Week 0) to the Study End (Week 362 ) and the Safety Follow-up (Week 372)
Population: All 310 subjects in the Safety Population are included in the analysis of this outcome measure. Safety Population includes all enrolled subjects who received at least one injection of study treatment in feeder study C87031 [NCT00152490] or C87032 [NCT00152425].
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 310
percentage of subjects | 94.2

2. Primary Outcome: Percentage of Subjects With at Least One Serious Adverse Event (SAE) During the Duration of This Study CDP870-034 (up to 84 Months)
Description: An SAE is defined as any untoward medical occurrence that occurs at any dose which results in death, is life threatening requires hospitalization, results in persistent/significant disability/incapacity, is an infection that requires parenteral antibiotics, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: Up to 84 months from Study Entry (Week 0) to the Study End (Week 362 ) and the Safety Follow-up (Week 372)
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 310
percentage of subjects | 44.5

3. Secondary Outcome: Percentage of Subjects Achieving Harvey Bradshaw Index (HBI) Remission (HBI ≤ 4) at Study Completion Visit or (Early) Withdrawal Visit
Description: HBI remission is defined as total HBI score of 4 points or less. HBI score consists of clinical parameters of general well-being (0 to 4), abdominal pain (0 to 3), number of liquid stools per day, abdominal mass (0 to 3), and complications (8 items, score 1 per item) lower scores indicating better well being. The first three parameters are scored for the previous day.
Time Frame: Study Completion Visit (Week 362) / (Early) Withdrawal Visit
Population: All 309 subjects in the Intention-To-Treat (ITT) Population are included in the analysis of this outcome measure. ITT Population includes all subjects of the Safety Population who provide at least one efficacy measurement after Week 0 of this study.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 309
percentage of subjects | 34.6 [29.3 to 39.9]

4. Secondary Outcome: Percentage of Subjects in Harvey Bradshaw Index (HBI) Response (HBI Change ≥ 3) at Study Completion Visit or (Early) Withdrawal Visit From Week 0 of Feeder Study CDP870-031 or CDP870-032
Description: Response is defined as decrease in total Harvey Bradshaw Index (HBI) score of 3 or more points. HBI score consists of clinical parameters of general well-being (0 to 4), abdominal pain (0 to 3), number of liquid stools per day, abdominal mass (0 to 3), and complications (8 items, score 1 per item) lower scores indicating better well being. The first three parameters are scored for the previous day.
Time Frame: From Baseline of study CDP870-031 [NCT00152490] or CDP870-032 [NCT00152425] to Study Completion Visit (Week 362) or (Early) Withdrawal Visit of this study (up to 90 months)
Population: Of the 309 subjects in the Intention-To-Treat (ITT) Population, 307 subjects are included in the analysis of this outcome measure. ITT Population includes all subjects of the Safety Population who provide at least one efficacy measurement after Week 0 of this study.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 307
percentage of subjects | 52.8 [47.2 to 58.4]

5. Secondary Outcome: Percentage of Subjects in Harvey Bradshaw Index (HBI) Response (HBI Change ≥ 3) at Study Completion Visit or (Early) Withdrawal Visit From Week 0 of CDP870-034
Description: as for outcome 4
Time Frame: From Week 0 of study CDP870-034 to Study Completion Visit (Week 362) or (Early) Withdrawal Visit (up to 84 months)
Population: Of the 309 subjects in the Intention-To-Treat (ITT) Population, 299 subjects are included in the analysis of this outcome measure. ITT Population includes all subjects of the Safety Population who provide at least one efficacy measurement after Week 0 of this study.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 299
percentage of subjects | 65.6 [60.2 to 70.9]

6. Secondary Outcome: Plasma Concentration of Certolizumab Pegol at Study Completion Visit or (Early) Withdrawal Visit
Description: Plasma Samples for determination of Certolizumab Pegol were taken prior to Certolizumab Pegol administration.
Time Frame: Study Completion Visit (Week 362) / (Early) Withdrawal Visit
Population: Of the 310 subjects in the Safety Population, 307 subjects are included in the analysis of this outcome measure. Safety Population includes all enrolled subjects who received at least one injection of study treatment in feeder study C87031 [NCT00152490] or C87032 [NCT00152425].
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 307
µg/mL | 5.870 [4.915 to 7.009]

7. Secondary Outcome: Percentage of Subjects With Positive Anti-CZP Anti-body Status at Any Time From Week 0 of the Feeder Studies CDP870-031 or CDP870-032 to the Study Completion Visit in CDP870-034
Description: Subjects are counted as antibody positive to Certolizumab Pegol if they have at least one positive result from Week 0 in one of the previous studies CDP870-031 [NCT00152490] or CDP870-032 [NCT00152425] to the last Visit in this study. A positive result is defined as Anti-CZP antibody levels > 2.4 units/mL.
Time Frame: From Week 0 of study CDP870-031 [NCT00152490] or CDP870-032 [NCT00152425] up to Study Completion Visit (Week 362) of CDP870-034 (up to 90 months)
Population: Of the 310 subjects in the Safety Population, 309 subjects are included in the analysis of this outcome measure. Safety Population includes all enrolled subjects who received at least one injection of study treatment in feeder study C87031 [NCT00152490] or C87032 [NCT00152425].
Measure: Number; unit: percentage of subjects
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 309
percentage of subjects | 23.6

8. Secondary Outcome: C-Reactive Protein (CRP) Level at Study Completion Visit or (Early) Withdrawal Visit
Time Frame: Study Completion Visit (Week 362) / (Early) Withdrawal Visit
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 309
mg/L | 10.78 [9.28 to 12.53]

9. Secondary Outcome: Fecal Calprotectin Level at Week 256 or (Early) Withdrawal Visit, if it is Earlier Than Week 256
Time Frame: Week 256 / (Early) Withdrawal Visit, if it is earlier than Week 256
Population: Of the 309 subjects in the Intention-To-Treat (ITT) Population, 280 subjects are included in the analysis of this outcome measure. ITT Population includes all subjects of the Safety Population who provide at least one efficacy measurement after Week 0 of this study.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/g stool
Arm/Group | Certolizumab Pegol
Number analyzed (Participants) | 280
µg/g stool | 460.784 [382.149 to 555.599]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected up to approximately 7 years, from Study Entry (Week 0) to the Safety Follow-up (Week 372).
Description: Adverse Events refer to the Safety Population, including all enrolled subjects who received at least one injection of study treatment in feeder study C87031 [NCT00152490] or C87032 [NCT00152425].
Arm/Group | Certolizumab Pegol
Serious Adverse Events (participants affected / at risk) | 138/310
Other Adverse Events (participants affected / at risk) | 248/310
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=310)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Secondary anaemia (Blood and lymphatic system disorders) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Pigmented naevus (Congenital, familial and genetic disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Optic neuritis (Eye disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 49 (50)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Small intestinal obstruction (Gastrointestinal disorders) | 7 (9)
Colonic stenosis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Ileal stenosis (Gastrointestinal disorders) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 2 (3)
Irritable bowel syndrome (Gastrointestinal disorders) | 2 (3)
Perirectal abscess (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Anal discomfort (Gastrointestinal disorders) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Gastroduodenitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal irritation (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Intestinal fistula (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Jejunal perforation (Gastrointestinal disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Rectal stenosis (Gastrointestinal disorders) | 1 (1)
Rectovaginal fistula (Gastrointestinal disorders) | 1 (1)
Small intestinal stricture (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Chest pain (General disorders) | 2 (2)
General physical health deterioration (General disorders) | 1 (1)
Impaired healing (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1)
Perianal abscess (Infections and infestations) | 9 (10)
Abdominal abscess (Infections and infestations) | 4 (4)
Sepsis (Infections and infestations) | 4 (4)
Abscess intestinal (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 2 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Anal fistula infection (Infections and infestations) | 1 (1)
Appendiceal abscess (Infections and infestations) | 1 (1)
Breast abscess (Infections and infestations) | 1 (1)
Bronchitis acute (Infections and infestations) | 1 (1)
Cystitis acute (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Genital abscess (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Mastitis (Infections and infestations) | 1 (1)
Pelvic abscess (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Tonsillitis streptococcal (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Medical device complication (Injury, poisoning and procedural complications) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1)
Postoperative haematoma (Injury, poisoning and procedural complications) | 1 (1)
Venom poisoning (Injury, poisoning and procedural complications) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Sperm analysis abnormal (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Pregnancy on oral contraceptive (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Alcoholism (Psychiatric disorders) | 1 (1)
Bipolar I Disorder (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1)
Psychological factor affecting medical condition (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 3 (4)
Nephrolithiasis (Renal and urinary disorders) | 3 (3)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Vesical fistula (Renal and urinary disorders) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1)
Endometrioma (Reproductive system and breast disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Refusal of treatment by patient (Social circumstances) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Certolizumab Pegol (N=310)
Anaemia (Blood and lymphatic system disorders) | 18 (23)
Crohn's disease (Gastrointestinal disorders) | 107 (138)
Abdominal pain (Gastrointestinal disorders) | 62 (98)
Diarrhoea (Gastrointestinal disorders) | 41 (61)
Nausea (Gastrointestinal disorders) | 40 (55)
Vomiting (Gastrointestinal disorders) | 32 (50)
Constipation (Gastrointestinal disorders) | 18 (24)
Anal fissure (Gastrointestinal disorders) | 17 (29)
Dyspepsia (Gastrointestinal disorders) | 17 (20)
Abdominal pain upper (Gastrointestinal disorders) | 16 (18)
Pyrexia (General disorders) | 32 (45)
Fatigue (General disorders) | 20 (24)
Influenza like illness (General disorders) | 17 (21)
Nasopharyngitis (Infections and infestations) | 44 (71)
Urinary tract infection (Infections and infestations) | 36 (60)
Influenza (Infections and infestations) | 34 (56)
Upper respiratory tract infection (Infections and infestations) | 34 (69)
Sinusitis (Infections and infestations) | 26 (45)
Gastroenteritis (Infections and infestations) | 18 (23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 49 (65)
Back pain (Musculoskeletal and connective tissue disorders) | 29 (38)
Headache (Nervous system disorders) | 48 (61)
Anxiety (Psychiatric disorders) | 19 (28)
Insomnia (Psychiatric disorders) | 19 (22)
Depression (Psychiatric disorders) | 18 (20)
Rash (Skin and subcutaneous tissue disorders) | 25 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days